CLINICAL TRIAL: NCT03175133
Title: Targeted Strength Training to Improve Gait in People With Multiple Sclerosis: a Feasibility Study
Brief Title: Strength Training to Improve Gait in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-2610
Record Dates: First submitted 2017-05-23; First posted 2017-06-05 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
Keywords: rehabilitation; physical therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Strength training (Experimental): Strength exercises for ankle PF, hip abduction, and trunk muscles. Exercises will be done in three standard positions of supine, sidelying, prone, seated, and standing. Exercises during the initial 4 weeks will be completed 2x week with supervision of a physical therapist and 2x week at home, for a total of 4x week. For the final 4 weeks of the intervention will be completed 1x week with supervision and 3x week at home.
  Interventions: Other: Strength exercise

INTERVENTIONS:
Other: Strength exercise — Strengthening exercises performed with physical therapist.

SUMMARY:
This study will pilot a strengthening intervention targeted to muscles found to be important to gait in people with multiple sclerosis (MS). Previous studies that have tried to strengthen leg and trunk muscles in people with MS have failed to improve walking ability consistently. The investigators think that is because strengthening exercises were not targeted to the correct muscle groups. For this study the investigators propose targeting muscle groups that they have found to be strong contributors to walking in a prior study. This is the first study to target these muscles, so the investigators propose doing a small trial to first evaluate the feasibility of the strength program and the outcomes. The investigators will measure strength and walking measures twice before and once after an 8-week strengthening intervention in a single group of 10 people with MS who are able to walk independently. The results of this study will help inform future, larger trials that could change the way strength training is conducted in people with MS.

ELIGIBILITY:
Inclusion Criteria:

1. People with MS,
2. Age 18-65,
3. A confirmed diagnosis of MS, and
4. Are ambulatory for 100m without an assistive device (EDDS 0-5.5), and
5. Have a gait speed measured by time to walk the 25-foot walk test of at least five seconds.

Exclusion Criteria:

1. Subjects are not ambulatory,
2. Subjects rely on a wheelchair,
3. Subjects cannot ambulate 100m (EDDS 6 or greater) without use of assistive devices, braces, or orthotics,
4. Walk the T25FW in less than five seconds,
5. Have lower extremity spasticity of 2 or greater on the Modified Ashworth Scale (MAS),
6. Have pain or other conditions that limit ambulation or ability to test muscle strength,
7. Cannot give consent,
8. Cannot follow simple directions,
9. Have had an exacerbation in the past month,
10. Have had changes to their drug therapy in the last month,
11. Have other neurologic diagnoses, or
12. Are currently undergoing physical therapy for strength training.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Strength | Week 0 (Baseline 1); Week 1 (Baseline 2); Week 10 (Follow-Up)
  Muscle strength measured by hand-held dynamometry (HHD) and clinical strength tests
Change in Timed 25 Foot Walk (T25FW) | Week 0 (Baseline 1); Week 1 (Baseline 2); Week 10 (Follow-Up)
  Gait speed over a 25 foot distance

SECONDARY OUTCOMES:
Change in 6-Minute Walk Test | Week 0 (Baseline 1); Week 1 (Baseline 2); Week 10 (Follow-Up)
  Gait endurance
Change in Dynamic Gait Index | Week 0 (Baseline 1); Week 1 (Baseline 2); Week 10 (Follow-Up)
  Balance during gait and other functional activities
Change in Multiple Sclerosis Walking Scale-12 | Week 0 (Baseline 1); Week 1 (Baseline 2); Week 10 (Follow-Up)
  Self-report measure of limitations in walking related activities
Change in Patient Specific Functional Scale | Week 0 (Baseline 1); Week 10 (Follow-Up)
  Self reported measure of self-selected limitations in participation

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Schenkman, PT, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manago MM, Hebert JR, Schenkman M. Psychometric Properties of a Clinical Strength Assessment Protocol in People with Multiple Sclerosis. Int J MS Care. 2017 Sep-Oct;19(5):253-262. doi: 10.7224/1537-2073.2016-078. PMID 29070966